CLINICAL TRIAL: NCT03982212
Title: A Window of Opportunity Trial of Intratumoral Injection of Copaxone® in Patients With Percutaneously Accessible Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-Copax-HN
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: Copaxone; Window of Opportunity Trial
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell | interventions — Glatiramer Acetate; Coat Protein Complex I

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, preoperative, window of opportunity trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intratumoral Copaxone (Experimental): Eligible subjects receive at least 1 and up to 3 doses of Copaxone® 40 milligrams (mg) intratumorally prior to standard of care surgery. The doses will be administered at least 48 hours apart. The last dose will be given within 96 hours of standard of care surgery.
  Interventions: Drug: Copaxone

INTERVENTIONS:
Drug: Copaxone — * Agent: Glatiramer acetate (Copaxone®)
  * Dose: 40 mg
  * Route: Intratumoral injection
  * Schedule: At least 1 dose, up to 3 doses, with each dose being at least 48 hours apart and last dose within 96 hours of standard of care surgery.
  Other Names: Glatiramer acetate; Glatopa

SUMMARY:
The investigator believes that injecting Copaxone into tumors will help participants immune system fight cancer. This has been studied in mice and has shown encouraging results. Copaxone is a safe medication currently used to treat Multiple Sclerosis (MS) and has very few side effects. To be considered for this trial a tumor must be easy to be injected and must be at least the size of a pea. Participants will be closely monitored for any side effects. Tissue from before surgery will be compared to tissue after the treatment and surgery to be checked for immune response and anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant or Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent.
* Have confirmed diagnosis of squamous cell cancer or cutaneous squamous cell cancer or basal cell carcinoma.
* Have one or more tumors measuring at least 5 mm in diameter.
* No prior therapy for this malignancy.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception (hormonal AND barrier method of birth control) prior to study entry, for the duration of study participation until the end of study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.
* Men of child-bearing potential must not father a child or donate sperm while on this study until the end of study treatment.
* Physician feels the patient is medically fit for the trial.

Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study.
* Pregnant or breast feeding. There is a potential for congenital abnormalities and for this regimen to harm breast feeding infants (if applicable) Planned treatment with chemotherapy and/or radiation therapy prior to standard of care surgery. Concurrent treatment with anti-cancer therapy is not allowed.
* Hypersensitivity to Copaxone® or glatiramer acetate, mannitol, or any component of the formulation.
* A known condition that leads to immunosuppression such as Acquired Immunodeficiency Syndrome (AIDS) or concurrent use of immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants that experience Treatment Related Adverse Events (TRAEs) or Treatment Related Serious Adverse Events (TRSAEs) | up to 6 weeks
  Participants will be evaluated for TRAEs and TRSAEs from the time of the first injection (Day 1) through the time they go to surgery. TRAEs and TRSAEs will be evaluated per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Immune Biomarker Level | Up to 6 weeks
  The Human V2 nCounter® Immunology Panel (NanoString Technologies) will be used to measure the difference of immune biomarker levels at pre-treatment and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquina Baranda, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (3):
- United States (3):
  - University of Kansas Cancer Center - CRC, Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baranda JC, Mohyuddin GR, Bur AM, Shnayder Y, Sweeney KR, Kakarala K, Prouty M, Pathak H, Puri R, Mitra A, Madan R, Forrest ML, Huang A, Weir S, Godwin AK, Alhakamy NA, Griffin JD, Berkland CJ. A window of opportunity trial evaluating intratumoral injection of Copaxone(R) in patients with percutaneously accessible tumors. Transl Med Commun. 2023;8:5. doi: 10.1186/s41231-023-00137-9. Epub 2023 Feb 27. PMID 40230575